CLINICAL TRIAL: NCT01281787
Title: Prevention of Atrial Fibrillation in Patients Undergoing Thoracic Surgery for Lung Cancer
Acronym: PRESAGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEO S365/407; 2007-003856-12 (EudraCT Number)
Record Dates: First submitted 2010-12-21; First posted 2011-01-24 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Lung Cancer; Atrial Fibrillation
Keywords: FAP= post-surgery atrial fibrillation; ACEI= angiotensin converting enzyme-inhibitors; ARBs= angiotensin II receptor blockers; NT-proBNP= brain natriuretic peptide
MeSH Terms: conditions — Lung Neoplasms; Atrial Fibrillation | interventions — Metoprolol; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Losartan (Active Comparator): angiotensin II-receptor blocker
  Interventions: Drug: Losartan
- no treatment (No Intervention): no preventive treatment
- Metoprolol (Active Comparator): beta-adrenergic antagonist
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Metoprolol — Metoprolol; 100 mg x 2 die (tablets); started within 12 hours after surgery and continued for the duration of hospital stay
  Other Names: SELOKEN, LOPRESOR
  Arms: Metoprolol
Drug: Losartan — Losartan; 50 mg die (tablets); started within 12 hours after surgery and continued for the duration of hospital stay
  Other Names: LORTAAN, NEOLOTAN, LOSAPREX
  Arms: Losartan

SUMMARY:
The aim of this study is to assess whether prophylactic treatment with metoprolol or losartan is able to reduce the incidence of atrial fibrillation (AF) in patients undergoing thoracic surgery for lung cancer, showing elevated plasma levels in NT probrain natriuretic peptide (NT-proBNP), measured in the perioperative period.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation is one of the most common complication after thoracic surgery for lung cancer, with an incidence ranging from 8 to 20% after lobectomy and up to 42% after pneumonectomy.

In a recent study we demonstrated that a high perioperative plasma levels of NT-proBNP is able to identify patients at risk for AF (incidence of 65%).

It has also been demonstrated that the renin-angiotensin system may play an important role in the pathophysiology of atrial fibrillation and that angiotensin converting enzyme inhibitors (ACEI) and angiotensin II receptor blockers (ARBs) are able to prevent atrial fibrillation in patients with heart failure, after myocardial infarction, in hypertensive patients and after electrical cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with age ≥ 18 years
* Thoracic surgery for lung cancer
* Evidence of elevated perioperative NT-proBNP
* Written informed consent

Exclusion Criteria:

* Hypersensitivity and / or intolerance to metoprolol or losartan
* History of heart failure
* Left ventricular ejection fraction <50% measured by echocardiographic techniques (Simpson rule)
* Permanent atrial fibrillation
* Antiarrhythmic therapy
* Current therapy with beta-blockers, angiotensin II receptor blockers and angiotensin-converting enzyme inhibitors
* Systolic blood pressure <95 mmHg
* Pregnant and lactating women

Additional exclusion criteria for therapy with beta-blocker:

* History of sick sinus syndrome, evidence of AV-block grade II or greater
* Heart rate <65 b / m
* History of bronchial asthma, severe bronchopneumopathy, evidence of bronchospasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2008-04; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative atrial fibrillation | up to 10 days

SECONDARY OUTCOMES:
Evaluation of NT-proBNP in the days following the start of treatment and post surgery duration of hospital stay | up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Cardinale, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Milan, Italy